CLINICAL TRIAL: NCT02672891
Title: Intrauterine Balloon Tamponade in the Management of Postpartum Hemorrhage in a Low Resource Setting
Brief Title: Intrauterine Balloon Tamponade in the Management of Postpartum Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia Obstetrics and Gynecology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MenoufiaOGG
Record Dates: First submitted 2015-12-23; First posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage; Uterine Tamponade; Condom Catheter
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device (Experimental): condom balloon catheter which is composed of a latex condom (SURE natural latex condom, Shanghai) and a 16-20 F, 2 ways silicon coated Foley catheter (Egypt). The catheter was introduced inside the condom and tied over tightly several times with a silk suture, to prevent air escape.
  Interventions: Device: condom balloon catheter

INTERVENTIONS:
Device: condom balloon catheter — The condom balloon catheters were inserted into the uterine cavity digitally or with forceps .Tight vaginal pack was inserted or cervical stitch was done to prevent displacement of the balloon catheter.
  (2)-Insertion at Cesarean Section: The catheter was inserted through the uterine incision (pushing the tip to the fundus and the drainage port through the cervix into the vagina) or transvaginally and inﬂated after the uterine incision was closed.

SUMMARY:
Intrauterine balloon tamponade in the management of postpartum hemorrhage in the obstetrics emergency ward in menoufiya university hospitals as a low resource setting.Guidelines for the management of postpartum hemorrhage involve a stepwise approach including the exclusion of retained products and genital tract trauma. Uterine atony, which is the most common cause, is dealt with uterine rubbing and various uterotonic agents. Among the new modalities introduced to arrest the bleeding is the uterine tamponade using various balloons and catheters. The condom catheter uses a sterile rubber catheter fitted with a condom for uterine tamponade .

DETAILED DESCRIPTION:
Objectives: To evaluate the outcome of uterine balloon tamponade using condom-catheter in the management of primary postpartum hemorrhage (PPH).

Material and Methods: Prospective observational study included 50 women with primary postpartum hemorrhage unresponsive to uterotonics and bimanual compression, was conducted at the department of Obstetrics &Gynecology, Menoufia University Hospital, Egypt. Clinical assessment, laboratory investigations and intrauterine condom catheter were applied to all patients. The primary outcome was the success of the balloon to stop bleeding, maternal complications were assessed as secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* women with primary postpartum hemorrhage ( defined as >500 ml estimated blood loss after vaginal delivery or >1000 ml after cesarean delivery)in the first 24 h , unresponsive to uterotonics and bimanual compression were enrolled

Exclusion Criteria:

* Patients with traumatic PPH, retained placenta, coagulopathy and severe systemic diseases were excluded from the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
control uterine bleeding (normal lochia). | 30 minutes

SECONDARY OUTCOMES:
Maternal complications (minor as fever and pain or major as blood transfusion, peripartum hysterectomy) | 24 hours
Maternal complications (admission to intensive care unit (ICU)) | 24 hours
Maternal complications (mortality) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hamed El Ellakwa, MD, Principal Investigator — Menoufiya faculty of medicine,menoufiya university,ministry of higher education
Locations (1):
- Menoufia University, Shebin Elkom, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes

REFERENCES:
- [Result] Schmidt J, Hotz HG, Foitzik T, Ryschich E, Buhr HJ, Warshaw AL, Herfarth C, Klar E. Intravenous contrast medium aggravates the impairment of pancreatic microcirculation in necrotizing pancreatitis in the rat. Ann Surg. 1995 Mar;221(3):257-64. doi: 10.1097/00000658-199503000-00007. PMID 7717779
- [Derived] Kandeel M, Sanad Z, Ellakwa H, El Halaby A, Rezk M, Saif I. Management of postpartum hemorrhage with intrauterine balloon tamponade using a condom catheter in an Egyptian setting. Int J Gynaecol Obstet. 2016 Dec;135(3):272-275. doi: 10.1016/j.ijgo.2016.06.018. Epub 2016 Aug 21. PMID 27599602